CLINICAL TRIAL: NCT01365156
Title: A Phase III Randomized Study of Pretherapeutic Para-aortic Lymphadenectomy in Women With Locally Advanced Cervical Cancer Dispositioned to Definitive Chemoradiotherapy
Brief Title: Extraperitoneal Para-aortic Lymph Node Dissection (EPLND) for Cervix
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0952; NCI-2011-02400 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Results first posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Cervical Squamous Cell Carcinoma; Adenosquamous Carcinoma; Adenocarcinoma; Locally Advanced Malignant Neoplasm; Cervical Cancer
Keywords: locally advanced cervical cancer; pretherapeutic para-aortic surgical staging; radiologic staging; pretherapeutic surgical staging; para-aortic metastatic disease
MeSH Terms: conditions — Carcinoma, Adenosquamous; Adenocarcinoma; Uterine Cervical Neoplasms | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EPLND + Chemoradiation (Experimental): Group 1: Extraperitoneal laparoscopic lymphadenectomy followed by chemoradiation therapy
  Interventions: Procedure: Extraperitoneal laparoscopic lymphadenectomy (EPLND); Radiation: Chemoradiation
- Chemoradiation (Active Comparator): Group 2: standard-of-care chemoradiation therapy only
  Interventions: Radiation: Chemoradiation

INTERVENTIONS:
Procedure: Extraperitoneal laparoscopic lymphadenectomy (EPLND) — Laparoscopic surgical procedure to remove and examine lymph nodes in abdomen, 7-10 days before chemoradiation treatment
  Other Names: Laparoscopic Extraperitoneal lymphadenectomy; Extraperitoneal Para-aortic Lymph Node Dissection; EPLND
  Arms: EPLND + Chemoradiation
Radiation: Chemoradiation — Radiation for 5 days in a row for 5 to 5½ weeks plus Cisplatin Chemotherapy cisplatin chemotherapy by vein over about 2 hours, 1 time every week for about 6 weeks.

SUMMARY:
The goal of this clinical research study is to learn if a surgical procedure called an extraperitoneal laparoscopic lymphadenectomy followed by chemotherapy and tailored radiation therapy can help to control the disease for a longer time than standard-of-care chemotherapy and whole pelvic radiation therapy.

DETAILED DESCRIPTION:
You will have a positron emission tomography/computed tomography (PET/CT) scan to check the status of the disease. For up to 6 hours before the PET/CT scan, you must not eat or drink anything except water. A small tube will be placed in your arm, and you will receive an injection of a very small amount of a mildly radioactive sugar material into your bloodstream. The radioactive nature of this injected material allows the scanner to "see" it in certain places in your body. After the injection, you will need to rest quietly until it is time for the scan. The amount of rest time may vary, but be prepared to wait for between 45 and 90 minutes. During the scan, you will lie flat on your back on a table. The scan itself may last up to 1 hour.

The study doctor will discuss the test results with you. If the test shows that you are not eligible to take part in the study, you will not be enrolled. Other treatment options will be discussed with you.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. You have an equal chance of being assigned to either group.

If you are in Group 1, you will have an extraperitoneal laparoscopic lymphadenectomy followed by chemoradiation therapy.

If you are in Group 2, you will receive standard-of-care chemoradiation therapy only.

Study Procedure and Visits:

If you are in Group 1, you will have an extraperitoneal laparoscopic lymphadenectomy, a procedure where surgeons remove and examine the lymph nodes in the abdomen. The study doctor will explain the risks for this procedure to you and you will sign a separate surgical consent form. This procedure will be performed 7-10 days before chemoradiation treatment begins.

During the laparoscopy procedure, a telescope-like instrument with a small camera on the end (a laparoscope) will be placed through a small cut in the abdomen. Three (3) other small cuts will be made to place instruments that may be needed to complete the surgery. Before the laparoscope is inserted, carbon dioxide gas will be pumped into your abdomen making it easier for the surgeon to see. The laparoscope will then be placed through the small cut. Using a TV monitor, the surgeon will use the camera to find the lymph nodes in the abdomen and then remove them. After the procedure is finished, the carbon dioxide gas will be removed and you will be taken to the recovery room.

If these lymph nodes contain cancer, the area of the body treated with radiation can be "extended" to treat new areas. Future treatment options will be based on what is found. This means that radiation will be used to treat both the lymph nodes in the abdomen and the standard area of radiation in the pelvis.

Participants in both groups will then have radiation for 5 days in a row for 5 to 5½ weeks. If the study doctor thinks it is needed and you agree, you will have extra radiation treatments.

Participants in both groups will receive cisplatin chemotherapy by vein over about 2 hours, 1 time every week for about 6 weeks. In most cases, treatment is given on Mondays (Days 1, 8, 15, 22, 29, and 36).

After 5 to 5½ weeks of chemotherapy and radiation treatment, participants in both groups will receive implants in the pelvis for about 48 hours. You will remain in the hospital at this time. The study doctor will explain the risks for this procedure to you and you will sign a separate surgical consent form.

Length of Study:

You may be on study for up to 5 years. Your participation on the study will be over after you have completed radiation treatment and the follow-up visits described below. You may be taken off study if intolerable side effects occur or if you are unable to follow study directions.

Long-Term Follow-Up:

The following tests and procedures will be performed:

* You will have a PET scan to check the status of the disease 3 months after you complete radiation treatment.
* You have a CT scan to check the status of the disease every 6 months for the next 3 years after that.

You will visit the clinic for a physical exam:

* Every 3 months for the first 2 years
* Every 6 months for the next 3 years, and
* One (1) time each year after that, up to 5 years

This is an investigational study. The extraperitoneal laparoscopic lymphadenectomy is considered investigational. Chemoradiation treatment is FDA approved for the treatment of cervical cancer.

Up to 600 patients will take part in this multicenter study. Up to 40 will be enrolled at MD Anderson. Up to 15 will be enrolled at the Harris Health System.

ELIGIBILITY:
Inclusion Criteria:

1. Women with clinical stage IB2-IVA cervical squamous cell carcinoma, adenosquamous, or adenocarcinoma.
2. Women with FDG-PET positive or indeterminate pelvic lymph nodes or indeterminate low common iliac nodes and negative paraaortic nodes.
3. Women with planned treatment of primary definitive chemoradiation therapy.
4. Patient information and written informed consent form signed.
5. Age >/= 18 years old
6. ECOG Performance Status (PS) </= 2
7. Life Expectancy >/= 3 months

Exclusion Criteria:

1. Women with stage IA or IB1 cancer.
2. Women with prior radiotherapy to the pelvis or retroperitoneal surgery.
3. Women with neuroendocrine histologies, or histologies other than squamous, adenosquamous or adenocarcinoma.
4. Women with FDG PETpositive high common or paraaortic lymph node metastasis confirmed by biopsy.
5. Women who have undergone simple or radical hysterectomy prior to radiotherapy.
6. Women with planned treatment of radiotherapy only (without chemotherapy).
7. Women with planned treatment of palliative radiotherapy.
8. Women with metastatic disease outside of pelvis.
9. Women who have completed treatment for other malignancies (except non-melanomatous skin cancer) < 5 years from their new diagnosis of cervical cancer.
10. Women who are pregnant, women who are likely to be pregnant or are breastfeeding.
11. Women with any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with patient's safety, provision of informed consent or compliance to study procedures.
12. (French Sites Only) Women not affiliated with Social Security System in France.
13. (French Sites Only) Women deprived of liberty or under guardianship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael M. Frumovitz, MD, MPH, Study Chair — M.D. Anderson Cancer Center
Locations (3):
- United States (2):
  - Lyndon B. Johnson General Hospital, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Vall d'Hebron Hospital, Brussels, Belgium

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 08/03/2011 and closed to new patient entry on 03/18/2016. All recruitments were done in a medical clinic setting.
Groups:
- Surgery Group: Laparoscopic extraperitoneal paraaortic lymphadenectomy followed by tailored chemoradiation
- Chemoradiation Group: Standard of care whole pelvic chemoradiation therapy
Period: Overall Study
Arm/Group | Surgery Group | Chemoradiation Group
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Surgery Group | Chemoradiation Group | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 47 [32 to 79] | 46 [25 to 60] | 46 [25 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 9 | 19
  Not Hispanic or Latino | 4 | 5 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 9 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  Spain | 4 | 4 | 8
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Rate
Description: To determine if patients with locally advanced cervical cancer have longer overall survivals with pretherapeutic paraaortic surgical staging followed by tailored chemoradiation when compared to patients who undergo standard radiologic staging followed by whole pelvic chemoradiation therapy.
Time Frame: 3 years
Population: Due to lack of funding and low accrual we were unable to determine the Overall Survival Rate.
Arm/Group | Surgery Group | Chemoradiation Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs will be collected from the time the patient signs the informed consent form up to 6 months post treatment, up to 8 years
Arm/Group | Surgery Group | Chemoradiation Group
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 5/14 | 3/14
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Surgery Group (N=14) | Chemoradiation Group (N=14)
Diarrhea (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Rectal Hemorrhage (Gastrointestinal disorders) | 1 | 1
Vaginal discharge (Reproductive system and breast disorders) | 1 | 1
Dyspareunia (Reproductive system and breast disorders) | 1 | 2
Hot flashes (Vascular disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-07-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT01365156/Prot_SAP_000.pdf